CLINICAL TRIAL: NCT06523062
Title: Short Term Reproducibility of Office White-coat Effect
Acronym: REBBRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 23-0196
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: White Coat Hypertension
Keywords: white coat effect; reproducibility; primary care
MeSH Terms: conditions — White Coat Hypertension | interventions — Blood Pressure Determination

STUDY DESIGN:
Intervention Model Description: cohort
Who Masked: Participant
Masking Description: adults > 18 y
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no reproducibility of OWCET (Other)
  Interventions: Device: blood pressure measurement
- reproducibility of OWCET (No Intervention)

INTERVENTIONS:
Device: blood pressure measurement — automated blood pressure measurement on 3 occasions at each consultation, twice with one month apart
  Arms: no reproducibility of OWCET

SUMMARY:
While a theoretical increase in systolic blood pressure (BP) of 10 mmHg can triple the relative risk of cardiovascular disease (CVD), the potential presence of a white coat effect (WCE) can interfere with the assessment of blood pressure control in the consultation. However, it is often difficult to assess the presence of a white coat effect (a quantitative variable) in general practice because of the difficulties in performing ambulatory BP measurements (self-measurement of blood pressure or ambulatory BP measurements). We have therefore previously described a surrogate concept of WCE obtained during a consultation with a general practitioner. It corresponds to a reduction of 10mmHg or more in systolic BP between the start and the end of the consultation. We have named it 'office white coat effect tail' (OWCET) and we have shown that OWCET, as a dichotomous variable, in a large Italian population cohort, with a follow-up of more than 18 years, was associated with an excess incidence of stroke, myocardial infarction (MI) and CVD and with excess mortality from MI and CVD. This concept appears to be more prevalent in women and is independent of blood pressure variability (regression to the mean). In addition, there is a genuine correlation between WCE and OWCET. To our knowledge, the reproducibility of the OWCET has never been studied, which could distort the relevance of this concept in the context of cardiovascular risk stratification in primary care.

ELIGIBILITY:
Inclusion Criteria:

* adult patients ;
* not taking any antihypertensive medication;
* free of any cardiovascular pathology.

Exclusion Criteria:

* patients who are minors or protected adults ;
* patients with BP ≥160/105 mmHg;
* history of secondary hypertension;
* taking a treatment that may affect blood pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 922 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
OWCET | 1 month
  Measurement of OWCET on two occasions during two consultations separated by one month, using the same automated blood pressure monitor, in order to estimate an intraclass kappa coefficient (qualitative measurement).

SECONDARY OUTCOMES:
Factors associated with reproducibility of OWCET | 1 month
  Patients characteristics
Different definitions of OWCET | 1 month
  Variation of OWCET definition in order to test OWCET reproducibility
blood pressure Variability | 1 month
  To test impact of blood pressure variability

IPD SHARING:
Plan to Share IPD: Yes
An initial inclusion visit, followed by a further visit at 1 month, with automated blood pressure measurement on 3 occasions at each visit, one month apart. At the first consultation, useful data were collected (age, sex, tobacco, alcohol, BMI, history of diabetes, history of chronic kidney disease, history of ischaemic heart disease).
Supporting Information: Study Protocol